CLINICAL TRIAL: NCT02872701
Title: A Phase 2, Single Dose, Open-Label, Exploratory Study to Investigate the Safety and Efficacy of OTL38 Injection for Intraoperative Imaging of Folate Receptor Positive Lung Nodules
Brief Title: OTL38 Injection for Intraoperative Imaging of Folate Receptor Positive Lung Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: On Target Laboratories, LLC (Industry)
Collaborators: Medelis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OTL-2016-OTL38-005
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Lung Neoplasms; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pafolacianine; Injections; Endoscopy; Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Patients Receiving OTL38 (Experimental): All patients in this arm will receive OTL38 for injection and undergo intraoperative imaging.
  Interventions: Drug: OTL38 for Injection; Device: Near infrared camera imaging system; Procedure: Endoscopic or Thoracic Surgery

INTERVENTIONS:
Drug: OTL38 for Injection — Folate analog ligand conjugated with an indole cyanine-like green dye as a solution in vials containing 3 mL at 2 mg/mL
  Other Names: OTL38
Device: Near infrared camera imaging system — Near infrared camera imaging system
Procedure: Endoscopic or Thoracic Surgery — Endoscopic or Thoracic Surgery

SUMMARY:
This is a phase 2, multi-center, single dose, open-label, exploratory study in suspected lung cancer patients scheduled to undergo endoscopic or thoracic surgery per CT/positron emission tomography imaging based on standard of care. This study aims to assess the efficacy of OTL38 and Near Infrared Imaging (NIR) at identifying pulmonary nodules within the operating theater, and to assess the safety and tolerability of single intravenous doses of OTL38.

DETAILED DESCRIPTION:
This is a phase 2, multi-center, single dose, open-label, exploratory study in suspected lung cancer patients scheduled to undergo endoscopic or thoracic surgery per CT/positron emission tomography (PET) imaging based on standard of care.

Two to three hours prior to surgery, patients will be infused with OTL38. After the patient is intubated and surgical site incised, the surgeon will locate and document all nodules identifiable by white light, manual palpation, and Near-Infrared Imaging (NIR). This will be documented and recorded. Surgery will be completed per surgeon's standard of care, afterwards the area will be reviewed under standard and infrared light. All samples will be sent for pathology and immunohistochemistry (IHC) evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients 18 years of age and older
2. Confirmed diagnosis of adenocarcinoma lung cancer OR,
3. Have a primary diagnosis, or at high clinical suspicion, of lung nodule(s) warranting surgery based on CT and/or PET imaging
4. Who are scheduled to undergo endoscopic or thoracic surgery surgery
5. A negative serum pregnancy test at Screening followed by a negative urine pregnancy test on the day of surgery or day of admission for female patients of childbearing potential
6. Female patients of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion
7. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

1. Previous exposure to OTL38
2. Known Folate Receptor-negative lung nodules
3. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient
4. History of anaphylactic reactions or severe allergies
5. History of allergy to any of the components of OTL38, including folic acid
6. Pregnancy, or positive pregnancy test
7. Clinically significant abnormalities on electrocardiogram (ECG) at screening.
8. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
9. Impaired renal function defined as epidermal growth factor receptor (eGFR) < 50 mL/min/1.73m2
10. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin.
11. Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to surgery
12. Known sensitivity to fluorescent light

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Receiving OTL38
Started | 100
Completed | 97
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 10
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity or True Positive Rate (TPR)
Description: Sensitivity or True Positive Rate (TPR) for OTL38 in combination with fluorescent light, defined as the proportion of fluorescent light positive tissue samples (nodule, synchronous lesion, and margin but excluding lymph nodes) that are histologically confirmed to be FR+ and lung cancer by central pathology relative to the total number of tissue samples confirmed to be FR+ and lung cancer by central pathology.
  Sensitivity = (True Positive)/(True Positive +False Negative)
Time Frame: 1 day
Population: The FAS for the analysis of the two co-primary endpoints, sensitivity and FPR, included patients exposed to OTL38 who:
  * Were evaluated under both normal light and fluorescent light imaging, and
  * Had central pathology and histology confirmation (positive for FR+ Lung Cancer) for at least one tissue sample detected under normal light or fluorescent light imaging
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: Lesions
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 107
proportion of lesions | 0.854 [0.74 to 0.92]

2. Primary Outcome: False Positive Rate (FPR)
Description: False positive rate (FPR) for OTL38 in combination with fluorescent light, for the purpose of this protocol, will be calculated as 1 - the Positive Predictive Value (PPV) and is defined as the proportion of fluorescent light positive tissue samples removed (nodule, synchronous lesion, and margin but excluding lymph nodes) that are histologically confirmed to be non-cancerous, or if cancerous, not FR+ and lung cancer, by central pathology relative to the total number of tissue samples removed with fluorescent light imaging. False Positive Rate = (False Positives) / (True Positives + False Positives)
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: Lesions
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 107
proportion of lesions | 0.138 [0.08 to 0.23]

3. Secondary Outcome: Proportion of Patients With at Least 1 Clinically Significant Event (CSE)
Description: Proportion of patients with at least 1 Clinically Significant Event (CSE as a result of utilizing OLT-38 and Near Infrared Imaging
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
proportion of participants | 0.293 [0.194 to 0.410]

4. Secondary Outcome: Positive Margin Identification
Description: Number of patients where at least one positive margin (fluorescent cancerous cells within 5 mm of the staple line) is identified with only OTL-38 and NIR
Time Frame: 1 day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
Participants | 8

5. Secondary Outcome: Synchronous Lesion Identification
Description: Number of patients where at least one synchronous lesions is identified only with OTL-38 and NIR
Time Frame: 1 day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
Participants | 7

6. Secondary Outcome: Pulmonary Nodule Identification
Description: Number of pulmonary nodules identified with OTL-38 and Near Infrared Imaging (NIR) that could not otherwise be identified by white light and palpation.
Time Frame: 1 day
Population: as for outcome 1
Measure: Number; unit: number of pulmonary nodules
Arm/Group | Patients Receiving OTL38
Number analyzed (Participants) | 75
number of pulmonary nodules | 10

ADVERSE EVENTS:
Time Frame: AEs were collected through Day 28 (+/- 4 days) from OTL38 administration
Arm/Group | Patients Receiving OTL38
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 14/100
Other Adverse Events (participants affected / at risk) | 94/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving OTL38 (N=100)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Arterial haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving OTL38 (N=100)
Procedural pain (Injury, poisoning and procedural complications) | 50 (50)
Incision site pain (Injury, poisoning and procedural complications) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 33 (33)
Vomiting (Gastrointestinal disorders) | 17 (17)
Constipation (Gastrointestinal disorders) | 10 (10)
Chest pain (General disorders) | 12 (12)
Fatigue (General disorders) | 10 (10)
Pyrexia (General disorders) | 6 (6)
Respiratory complication associated with device (General disorders) | 6 (6)
Hypertension (Vascular disorders) | 11 (11)
Hypotension (Vascular disorders) | 11 (11)
Atrial fibrillation (Cardiac disorders) | 8 (8)
Tachycardia (Cardiac disorders) | 5 (5)
Dizziness (Nervous system disorders) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Pneumonia (Infections and infestations) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02872701/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02872701/SAP_001.pdf